CLINICAL TRIAL: NCT02540993
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Event-driven Phase 3 Study to Investigate the Safety and Efficacy of Finerenone, in Addition to Standard of Care, on the Progression of Kidney Disease in Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Kidney Disease
Brief Title: Efficacy and Safety of Finerenone in Subjects With Type 2 Diabetes Mellitus and Diabetic Kidney Disease
Acronym: FIDELIO-DKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16244; 2015-000990-11 (EudraCT Number)
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Disease
Keywords: CKD; Diabetic Kidney Disease; Type 2 Diabetes; Kidney diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Diabetes Mellitus, Type 2; Kidney Diseases | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Finerenone (BAY94-8862) (Experimental): Participants received finerenone 10 mg or 20 mg once daily in addition to standard of care therapy
  Interventions: Drug: Finerenone (BAY94-8862)
- Placebo (Placebo Comparator): Participants received matching placebo once daily in addition to standard of care therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — Oral tablet; starting dose at 10 mg for subjects with an eGFR between 25 to < 60 mL/min/1.73m² at the Screening Visit; starting dose at 20 mg for subjects with an eGFR ≥ 60 mL/min/1.73m² at the Screening Visit; dose could be up-titrated from Month 1 onwards or down-titrated at any time during the study; once daily in the morning, until the trial was completed provided there were no safety grounds for discontinuing treatment
  Arms: Finerenone (BAY94-8862)
Drug: Placebo — Matching placebo, oral tablet, once daily in the morning, until the trial was completed provided there were no safety grounds for discontinuing treatment
  Arms: Placebo

SUMMARY:
The primary objective of this study was to demonstrate whether, in addition to standard of care, finerenone is superior to placebo in delaying the progression of kidney disease, as measured by the composite endpoint of time to first occurrence of kidney failure, a sustained decrease of estimated glomerular filtration rate (eGFR) ≥40% from baseline over at least 4 weeks, or renal death.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age
* Type 2 diabetes mellitus (T2D) as defined by the American Diabetes Association
* Diagnosis of chronic kidney disease (CKD) with at least one of the following criteria at run-in and screening visits:

  * persistent high albuminuria (UACR ≥30 to <300 mg/g in 2 out of 3 first morning void samples) and estimated glomerular filtration rate (eGFR) ≥25 but <60 mL/min/1.73 m² (CKD EPI) and presence of diabetic retinopathy or
  * persistent very high albuminuria (UACR ≥300 mg/g in 2 out of 3 first morning void samples) and eGFR ≥25 to <75 mL/min/1.73 m² (CKD-EPI)
* Prior treatment with angiotensin-converting enzyme inhibitors (ACEIs) and angiotensin receptor blockers (ARBs) as follows:

  * For at least 4 weeks prior to the run-in visit, subjects should be treated with either an ACEI or ARB, or both
  * Starting with the run-in visit, subjects should be treated with only an ACEI or ARB
  * For at least 4 weeks prior to the screening visit, subjects should be treated with the maximum tolerated labeled dose (but not below the minimal labeled dose) of only an ACEI or an ARB (not both) preferably without any adjustments to dose or choice of agent or to any other antihypertensive or antiglycemic treatment
* Serum potassium ≤4.8 mmol/L at both the run-in and the screening visit

Exclusion Criteria:

* Known significant non-diabetic renal disease, including clinically relevant renal artery stenosis
* Uncontrolled arterial hypertension (ie, mean sitting systolic blood pressure (SBP) ≥170 mmHg, sitting diastolic blood pressure (DBP) ≥110 mmHg at run-in visit, or mean sitting SBP ≥160 mmHg, sitting DBP ≥100 mmHg at screening)
* Glycated hemoglobin (HbA1c) >12%
* Mean SBP < 90 mmHg at the run-in visit or at the screening visit
* Clinical diagnosis of chronic heart failure with reduced ejection fraction (HFrEF) and persistent symptoms (New York Heart Association [NYHA] class II - IV) at run-in visit (class 1A recommendation for mineralcorticoid receptor antagonists [MRAs])
* Stroke, transient ischemic cerebral attack, acute coronary syndrome, or hospitalization for worsening heart failure, in the last 30 days prior to the screening visit
* Dialysis for acute renal failure within 12 weeks of run-in visit
* Renal allograft in place or scheduled within next 12 months from the run-in visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5734 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (707):
- United States (128):
  - Birmingham, Alabama
  - Fort Payne, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Prescott, Arizona
  - Tucson, Arizona
  - Arvin, California
  - Chula Vista, California
  - Dublin, California
  - El Centro, California
  - Fresno, California
  - La Mesa, California
  - Loma Linda, California
  - Los Angeles, California
  - Northridge, California
  - Port Hueneme, California
  - Poway, California
  - Rancho Cucamonga, California
  - Rialto, California
  - Roseville, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - New Haven, Connecticut
  - Waterbury, Connecticut
  - Fleming Island, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Gardens, Florida
  - Miami Lakes, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Duluth, Georgia
  - Lilburn, Georgia
  - Macon, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Elgin, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Hutchinson, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Metairie, Louisiana
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Flushing, New York
  - Mineola, New York
  - New York, New York
  - Rosedale, New York
  - Smithtown, New York
  - Staten Island, New York
  - Asheboro, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Beaver, Pennsylvania
  - Bethlehem, Pennsylvania
  - Hershey, Pennsylvania
  - Lansdale, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Murrells Inlet, South Carolina
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Kingwood, Texas
  - McAllen, Texas
  - McKinney, Texas
  - Pearland, Texas
  - Pflugerville, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - St. George, Utah
  - Burlington, Vermont
  - Alexandria, Virginia
  - Manassas, Virginia
  - Salem, Virginia
  - Virginia Beach, Virginia
  - Spokane Valley, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Argentina (9):
  - Junín, Buenos Aires
  - Lanús, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Sarandí, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - CABA, Ciudad Auton. de Buenos Aires
  - Ciudad Autón. de Buenos Aires, Ciudad Auton. de Buenos Aires
  - Córdoba
  - San Luis
- Australia (13):
  - Garran, Australian Capital Territory
  - Gosford, New South Wales
  - Liverpool, New South Wales
  - New Lambton, New South Wales
  - Wollongong, New South Wales
  - Adelaide, South Australia
  - Fitzroy, Victoria
  - Heidelberg, Victoria
  - Reservoir, Victoria
  - Richmond, Victoria
  - St Albans, Victoria
  - Box Hill
  - Elizabeth Vale
- Austria (9):
  - Graz, Styria
  - Saint Stefan, Styria
  - Linz, Upper Austria
  - Feldkirch, Vorarlberg
  - Innsbruck
  - Salzburg
  - Sankt Pölten
  - Vienna
  - Wels
- Belgium (9):
  - Antwerp
  - Bruxelles - Brussel
  - Edegem
  - Ghent
  - Ieper
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
- Brazil (17):
  - Fortaleza, Ceará
  - Feira de Santana, Estado de Bahia
  - Salvador, Estado de Bahia
  - Brasília, Federal District
  - Aparecida de Goiânia, Goiás
  - Goiânia, Goiás
  - Juiz de Fora, Minas Gerais
  - Curitiba, Paraná
  - Paraná, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - São José dos Campos, São Paulo
  - São Paulo, São Paulo
  - Minas Gerais
  - Rio de Janeiro
  - São Paulo
- Bulgaria (15):
  - Blagoevgrad
  - Botevgrad
  - Dimitrovgrad
  - Gorna Oryahovitsa
  - Kazanlak
  - Kozloduy
  - Lukovit
  - Plovdiv
  - Razgrad
  - Sliven
  - Smolyan
  - Sofia
  - Stara Zagora
  - Varna
  - Yambol
- Canada (23):
  - Burnaby, British Columbia
  - Coquitlam, British Columbia
  - New Westminster, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Smith Falls, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Greenfield Park, Quebec
  - Laval, Quebec
  - Mirabel, Quebec
  - Montreal, Quebec
  - Québec
- Chile (6):
  - Osorno, Los Lagos Region
  - Las Condes, Santiago Metropolitan
  - Providencia, Santiago Metropolitan
  - San Bernardo, Santiago Metropolitan
  - San Miguel, Santiago Metropolitan
  - Santiago
- China (31):
  - Fuzhou, Fujian
  - Xiamen, Fujian
  - Lanzhou, Gansu
  - Guangzhou, Guangdong
  - Zhuhai, Guangdong
  - Nanning, Guangxi
  - Haikou, Hainan
  - Wuhan, Hubei
  - Changsha, Hunan
  - Changzhou, Jiangsu
  - Huai'an, Jiangsu
  - Lianyungang, Jiangsu
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Wuxi, Jiangsu
  - Yancheng, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shenyang, Liaoning
  - Yinchuan, Ningxia
  - Xi'an, Shaanxi
  - Qingdao, Shandong
  - Taiyuan, Shanxi
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Taizhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Colombia (11):
  - Medellín, Antioquia
  - Baranquilla, Atlántico
  - Barranquilla, Atlántico
  - Bogotá, Bogota D.C.
  - Cundinamarca, Bogota D.C.
  - Manizales, Caldas Department
  - Zipaquirá, Cundinamarca
  - Armenia, Quindío Department
  - Cali, Valle del Cauca Department
  - Floridablanca
  - Medellín
- Czechia (17):
  - Beroun
  - Brandýs nad Labem
  - Břeclav
  - Česká Lípa
  - Český Krumlov
  - Frýdek-Místek
  - Hodonín
  - Holešov
  - Hranice
  - Kopřivnice
  - Krnov
  - Mladá Boleslav
  - Olomouc
  - Ostrava
  - Pilsen
  - Prague
  - Vlašim
- Denmark (14):
  - Aalborg
  - Aarhus N
  - Esbjerg
  - Hellerup
  - Herlev
  - Hillerød
  - Holbæk
  - Holstebro
  - Hvidovre
  - Kolding
  - København NV
  - Odense C
  - Svendborg
  - Viborg
- Finland (12):
  - Jyväskylä
  - Kajaani
  - Kerava
  - Klaukkala
  - Kuopio
  - Nurmijärvi
  - Oulu
  - Rauma
  - Seinäjoki
  - Tampere
  - Turku
  - Vantaa
- France (20):
  - Bois-Guillaume
  - Bordeaux
  - Boulogne-sur-Mer
  - Brest
  - Colmar
  - Dijon
  - La Rochelle
  - La Tronche
  - Le Coudray
  - Le Creusot
  - Lyon
  - Mulhouse
  - Nîmes
  - Paris
  - Pessac
  - Saint-Herblain
  - Saint-Priest-en-Jarez
  - Tourcoing
  - Vandœuvre-lès-Nancy
  - Vénissieux
- Germany (26):
  - Heidelberg, Baden-Wurttemberg
  - Ludwigsburg, Baden-Wurttemberg
  - Schweinfurt, Bavaria
  - Würzburg, Bavaria
  - Elsterwerda, Brandenburg
  - Bad König, Hesse
  - Frankfurt am Main, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Bad Oeynhausen, North Rhine-Westphalia
  - Bochum, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Nettetal, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Hoyerswerda, Saxony
  - Leipzig, Saxony
  - Jena, Thuringia
  - Berlin
  - Hamburg
- Greece (6):
  - Alexandroupoli
  - Athens
  - Chaïdári
  - Larissa
  - Nea Ionia
  - Thessaloniki
- Hong Kong (4):
  - Hong Kong
  - Shatin
  - Sheung Wan
  - Wong Tai Sin
- Hungary (14):
  - Baja
  - Balatonfüred
  - Budapest
  - Debrecen
  - Eger
  - Kistarcsa
  - Nyíregyháza
  - Pápa
  - Siófok
  - Szeged
  - Szentes
  - Székesfehérvár
  - Szombathely
  - Veszprém
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Israel (17):
  - Afula
  - Ashkelon
  - Beersheba
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Ramat Gan
  - Rehovot
  - Safed
  - Sakhnin
  - Tel Aviv
  - Tiberias
  - Ẕerifin
- Italy (15):
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Monza Brianza, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Messina, Sicily
  - Padua, Veneto
  - Verona, Veneto
- Japan (49):
  - Nagoya, Aichi-ken
  - Toyota, Aichi-ken
  - Funabashi, Chiba
  - Ichikawa, Chiba
  - Matsuyama, Ehime
  - Chikushino-shi, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Shirakawa, Fukushima
  - Ōgaki, Gifu
  - Maebashi, Gunma
  - Higashihiroshima, Hiroshima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Obihiro, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Naka, Ibaraki
  - Ushiku, Ibaraki
  - Komatsu, Ishikawa-ken
  - Sanuki, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Atsugi, Kanagawa
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Yokohama, Kanagawa
  - Tamana, Kumamoto
  - Yatsushiro, Kumamoto
  - Sasebo, Nagasaki
  - Beppu, Oita Prefecture
  - Yufu, Oita Prefecture
  - Nakagami-gun, Okinawa
  - Shimajiri, Okinawa
  - Suita, Osaka
  - Kawaguchi, Saitama
  - Sayama, Saitama
  - Ōtsu, Shiga
  - Iwata, Shizuoka
  - Oyama, Tochigi
  - Minato, Tokyo
  - Musashino, Tokyo
  - Shibuya-ku, Tokyo
  - Fukui
  - Fukuoka
  - Kagoshima
  - Kumamoto
  - Nagasaki
  - Osaka
  - Saitama
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Utena
  - Vilnius
- Malaysia (8):
  - Johor Bahru
  - Kelantan
  - Kuala Lumpur
  - Kuala Pahang
  - Kuala Selangor
  - Perak
  - Pulau Pinang
  - Putrajaya
- Mexico (14):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - México D.F., Mexico City
  - México, D. F., Mexico City
  - Cuernavaca, Morelos
  - Querétaro City, Querétaro
  - San Juan del Río, Querétaro
  - Culiacán, Sinaloa
  - Mazatlán, Sinaloa
  - Puerto de Veracruz, Veracruz
  - Xalapa, Veracruz
  - Aguascalientes
  - Chihuahua City
  - Mexico City
- Netherlands (14):
  - Alkmaar
  - Almere Stad
  - Amersfoort
  - Amsterdam
  - Apeldoorn
  - Breda
  - Dordrecht
  - Eindhoven
  - Geleen
  - Groningen
  - Hoogeveen
  - Nieuwegein
  - The Hague
  - Zwijndrecht
- New Zealand (7):
  - Auckland
  - Christchurch
  - Hamilton
  - Hawkes Bay
  - Palmerston North
  - Tauranga
  - Wellington
- Norway (8):
  - Ålesund
  - Hamar
  - Kløfta
  - Kristiansand
  - Levanger
  - Oslo
  - Skedsmokorset
  - Trondheim
- Philippines (4):
  - Iloilo City
  - Marikina City
  - Pasig
  - Quezon City
- Poland (18):
  - Bialystok
  - Bydgoszcz
  - Chojnice
  - Gdansk
  - Gdynia
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Poznan
  - Rzeszów
  - Skorzewo
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
  - Zabrze
- Portugal (14):
  - Covilha, Castelo Branco District
  - Loures, Lisbon District
  - Funchal, Madeira
  - Matosinhos Municipality, Porto District
  - Torres Novas, Santarém District
  - Setúbal, Setúbal District
  - Almada
  - Amadora
  - Braga
  - Faro
  - Leiria
  - Lisbon
  - Porto
  - Viana do Castelo
- Puerto Rico (2):
  - Cidra
  - San Juan
- Romania (11):
  - Alba Iulia, Alba
  - Baia Mare, Maramureş
  - Ploieşti, Prahova
  - Timișoara, Timiș County
  - Bucharest
  - Cluj-Napoca
  - Galati
  - Iași
  - Oradea
  - Satu Mare
  - Timișoara
- Russia (25):
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Irkutsk
  - Izhevsk
  - Kazan'
  - Kemerovo
  - Kirov
  - Krasnodar
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Orenburg
  - Perm
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Stavropol
  - Syktyvkar
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Singapore, Singapore
- Slovakia (5):
  - Bardejov
  - Nitra
  - Rimavská Sobota
  - Rožňava
  - Žilina
- South Africa (17):
  - Port Elizabeth, Eastern Cape
  - Benoni, Gauteng
  - Johannesburg, Gauteng
  - Lenasia South, Gauteng
  - Newtown, Gauteng
  - Petoria, Gauteng
  - Pretoria, Gauteng
  - Soweto, Gauteng
  - Durban, KwaZulu-Natal
  - Isipingo Rail, KwaZulu-Natal
  - Tongaat, KwaZulu-Natal
  - Middelburg, Mpumalanga
  - Witbank, Mpumalanga
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
  - Pretoria
- South Korea (9):
  - Chuncheon, Gang''weondo
  - Wŏnju, Gang''weondo
  - Anyang-si, Gyeonggido
  - Goyang-si, Gyeonggido
  - Incheon Gwangyeogsi,, Incheon Gwang''yeogsi
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daejeon
  - Seoul
- Spain (18):
  - Ferrol, A Coruña
  - Badalona, Barcelona
  - Manresa, Barcelona
  - Sant Joan Despí, Barcelona
  - Jerez de la Frontera, Cádiz
  - Burela de Cabo, Lugo
  - Alcalá de Henares, Madrid
  - Boadilla del Monte, Madrid
  - Getafe, Madrid
  - Sagunto, Valencia
  - A Coruña
  - Barcelona
  - Córdoba
  - Granada
  - Jaén
  - Madrid
  - Málaga
  - Valencia
- Sweden (7):
  - Gothenburg
  - Lund
  - Örebro
  - Rättvik
  - Skövde
  - Stockholm
  - Uppsala
- Switzerland (7):
  - Liestal, Basel-Landschaft
  - Geneva, Canton of Geneva
  - Olten, Canton of Solothurn
  - Sankt Gallen, Canton of St. Gallen
  - Lausanne, Canton of Vaud
  - Frauenfeld, Thurgau
  - Bern
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Turkey (Türkiye) (9):
  - Ankara
  - Antalya
  - Edirne
  - Izmir
  - Kayseri
  - Kocaeli
  - Malatya
  - Samsun
  - Sivas
- Ukraine (13):
  - Cherkasy
  - Chernivtsi
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Mykolayiv
  - Ternopil
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (13):
  - Llanelli, Carmarthenshire
  - Leicester, Leicestershire
  - Salford, Manchester
  - Liverpool, Merseyside
  - Northampton, Northamptonshire
  - Carshalton, Surrey
  - Newcastle upon Tyne, Vale of Glamorgan, the
  - Chichester, West Sussex
  - Bristol
  - London
  - Manchester
  - Middlesbrough
  - Portsmouth
- Vietnam (2):
  - Hà Nội
  - Ho Chi Minh City

REFERENCES:
- [Background] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Nowack C, Kolkhof P, Ferreira AC, Schloemer P, Filippatos G; on behalf of the FIDELIO-DKD study investigators; FIDELIO-DKD study investigators. Design and Baseline Characteristics of the Finerenone in Reducing Kidney Failure and Disease Progression in Diabetic Kidney Disease Trial. Am J Nephrol. 2019;50(5):333-344. doi: 10.1159/000503713. Epub 2019 Oct 25. PMID 31655812
- [Result] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825
- [Result] Filippatos G, Anker SD, Agarwal R, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Schloemer P, Tornus I, Joseph A, Bakris GL; FIDELIO-DKD Investigators. Finerenone and Cardiovascular Outcomes in Patients With Chronic Kidney Disease and Type 2 Diabetes. Circulation. 2021 Feb 9;143(6):540-552. doi: 10.1161/CIRCULATIONAHA.120.051898. Epub 2020 Nov 16. PMID 33198491
- [Derived] Mendoza JM, Weir MR, Anker SD, Filippatos G, Rossing P, Ahlers C, Brinker M, Fatoba ST, Horvat-Broecker A, Rohwedder K, Fornoni A; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone in People with CKD, Type 2 Diabetes, and History of Nephrectomy. Clin J Am Soc Nephrol. 2026 Jan 14. doi: 10.2215/CJN.0000000932. Online ahead of print. No abstract available. PMID 41533467
- [Derived] Katayama S, Anker SD, Zhu D, Kim S, Wu MJ, Kawanami D, Rossing P, Ruilope LM, Ahlers C, Brinker M, Mann A, Tian Y, Yamashita S, Pitt B; FIDELIO-DKD and FIGARO-DKD Investigators. Efficacy and safety of finerenone in Asian patients with type 2 diabetes and chronic kidney disease: A FIDELITY analysis by baseline kidney function. J Diabetes Complications. 2026 Jan;40(1):109213. doi: 10.1016/j.jdiacomp.2025.109213. Epub 2025 Nov 4. PMID 41289823
- [Derived] Mottl A, Scott C, Green JB, Heerspink HJL, Mann JFE, McGill JB, Nangaku M, Rosenstock J, Rossing P, Li L, Li N, Vaduganathan M, Agarwal R; CONFIDENCE Trial Investigators. Baseline Kidney Function, Albuminuria, and Urine Albumin-Creatinine Ratio Reduction with Finerenone, Empagliflozin, or Both: Post Hoc Analyses of CONFIDENCE Trial. J Am Soc Nephrol. 2025 Nov 6. doi: 10.1681/ASN.0000000928. Online ahead of print. No abstract available. PMID 41196655
- [Derived] Ferreira JP, Mendonca L, Marques P, Neves JS, Zannad F, Packer M. Albuminuria Is the Key Driver of Kidney Benefit with Aldosterone Receptor Antagonists in Type 2 Diabetes. J Am Soc Nephrol. 2025 Sep 2. doi: 10.1681/ASN.0000000877. Online ahead of print. No abstract available. PMID 40892478
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] Rossing P, Birkenfeld AL, Fioretto P, McGill JB, Anker SD, Pitt B, Rohwedder K, Scalise A, Scott C, Filippatos G; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone and Clinical Outcomes in CKD and Type 2 Diabetes by Frailty Index: FIDELITY Post Hoc Analysis. Clin J Am Soc Nephrol. 2025 May 2;20(7):968-977. doi: 10.2215/CJN.0000000700. PMID 40315020
- [Derived] Pitt B, Agarwal R, Anker SD, Rossing P, Ruilope L, Herzog CA, Greenberg B, Pecoits-Filho R, Lambelet M, Lawatscheck R, Scalise A, Filippatos G. Hypokalaemia in patients with type 2 diabetes and chronic kidney disease: the effect of finerenone-a FIDELITY analysis. Eur Heart J Cardiovasc Pharmacother. 2025 Feb 8;11(1):10-19. doi: 10.1093/ehjcvp/pvae074. PMID 39380152
- [Derived] Bansal S, Canziani MEF, Birne R, Anker SD, Bakris GL, Filippatos G, Rossing P, Ruilope LM, Farjat AE, Kolkhof P, Lage A, Brinker M, Pitt B. Finerenone cardiovascular and kidney outcomes by age and sex: FIDELITY post hoc analysis of two phase 3, multicentre, double-blind trials. BMJ Open. 2024 Mar 19;14(3):e076444. doi: 10.1136/bmjopen-2023-076444. PMID 38508632
- [Derived] Agarwal R, Tu W, Farjat AE, Farag YMK, Toto R, Kaul S, Lawatscheck R, Rohwedder K, Ruilope LM, Rossing P, Pitt B, Filippatos G, Anker SD, Bakris GL; FIDELIO-DKD and FIGARO-DKD Investigators. Impact of Finerenone-Induced Albuminuria Reduction on Chronic Kidney Disease Outcomes in Type 2 Diabetes : A Mediation Analysis. Ann Intern Med. 2023 Dec;176(12):1606-1616. doi: 10.7326/M23-1023. Epub 2023 Dec 5. PMID 38048573
- [Derived] Flack JM, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Adler SG, Fried L, Jamerson K, Toto R, Brinker M, Farjat AE, Kolkhof P, Lawatscheck R, Joseph A, Bakris GL; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone in Black Patients With Type 2 Diabetes and CKD: A Post hoc Analysis of the Pooled FIDELIO-DKD and FIGARO-DKD Trials. Kidney Med. 2023 Sep 28;5(12):100730. doi: 10.1016/j.xkme.2023.100730. eCollection 2023 Dec. PMID 38046911
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Rosas SE, Ruilope LM, Anker SD, Pitt B, Rossing P, Bonfanti AAC, Correa-Rotter R, Gonzalez F, Munoz CFJ, Pergola P, Umpierrez GE, Scalise A, Scott C, Lawatscheck R, Joseph A, Bakris GL; FIDELIO-DKD and FIGARO-DKD investigators. Finerenone in Hispanic Patients With CKD and Type 2 Diabetes: A Post Hoc FIDELITY Analysis. Kidney Med. 2023 Aug 1;5(10):100704. doi: 10.1016/j.xkme.2023.100704. eCollection 2023 Oct. PMID 37745646
- [Derived] Sarafidis P, Agarwal R, Pitt B, Wanner C, Filippatos G, Boletis J, Tuttle KR, Ruilope LM, Rossing P, Toto R, Anker SD, Liu ZH, Joseph A, Ahlers C, Brinker M, Lawatscheck R, Bakris G; FIDELIO-DKD and FIGARO-DKD Investigators. Outcomes with Finerenone in Participants with Stage 4 CKD and Type 2 Diabetes: A FIDELITY Subgroup Analysis. Clin J Am Soc Nephrol. 2023 May 1;18(5):602-612. doi: 10.2215/CJN.0000000000000149. Epub 2023 Apr 7. PMID 36927680
- [Derived] Agarwal R, Pitt B, Palmer BF, Kovesdy CP, Burgess E, Filippatos G, Malyszko J, Ruilope LM, Rossignol P, Rossing P, Pecoits-Filho R, Anker SD, Joseph A, Lawatscheck R, Wilson D, Gebel M, Bakris GL. A comparative post hoc analysis of finerenone and spironolactone in resistant hypertension in moderate-to-advanced chronic kidney disease. Clin Kidney J. 2022 Oct 30;16(2):293-302. doi: 10.1093/ckj/sfac234. eCollection 2023 Feb. PMID 36864892
- [Derived] Filippatos G, Anker SD, August P, Coats AJS, Januzzi JL, Mankovsky B, Rossing P, Ruilope LM, Pitt B, Sarafidis P, Teerlink JR, Kapelios CJ, Gebel M, Brinker M, Joseph A, Lage A, Bakris G, Agarwal R. Finerenone and effects on mortality in chronic kidney disease and type 2 diabetes: a FIDELITY analysis. Eur Heart J Cardiovasc Pharmacother. 2023 Feb 2;9(2):183-191. doi: 10.1093/ehjcvp/pvad001. PMID 36639130
- [Derived] Filippatos G, Anker SD, Pitt B, Rossing P, Joseph A, Kolkhof P, Lambelet M, Lawatscheck R, Bakris GL, Ruilope LM, Agarwal R. Finerenone and Heart Failure Outcomes by Kidney Function/Albuminuria in Chronic Kidney Disease and Diabetes. JACC Heart Fail. 2022 Nov;10(11):860-870. doi: 10.1016/j.jchf.2022.07.013. Epub 2022 Oct 12. PMID 36328655
- [Derived] Pitt B, Agarwal R, Anker SD, Ruilope LM, Rossing P, Ahlers C, Brinker M, Joseph A, Lambelet M, Lawatscheck R, Filippatos GS; FIDELIO-DKD and FIGARO-DKD Investigators. Association of Finerenone Use With Reduction in Treatment-Emergent Pneumonia and COVID-19 Adverse Events Among Patients With Type 2 Diabetes and Chronic Kidney Disease: A FIDELITY Pooled Secondary Analysis. JAMA Netw Open. 2022 Oct 3;5(10):e2236123. doi: 10.1001/jamanetworkopen.2022.36123. PMID 36287567
- [Derived] Ruilope LM, Agarwal R, Anker SD, Filippatos G, Pitt B, Rossing P, Sarafidis P, Schmieder RE, Joseph A, Rethemeier N, Nowack C, Bakris GL; FIDELIO-DKD Investigators. Blood Pressure and Cardiorenal Outcomes With Finerenone in Chronic Kidney Disease in Type 2 Diabetes. Hypertension. 2022 Dec;79(12):2685-2695. doi: 10.1161/HYPERTENSIONAHA.122.19744. Epub 2022 Oct 12. PMID 36252131
- [Derived] Filippatos G, Anker SD, Pitt B, McGuire DK, Rossing P, Ruilope LM, Butler J, Jankowska EA, Michos ED, Farmakis D, Farjat AE, Kolkhof P, Scalise A, Joseph A, Bakris GL, Agarwal R. Finerenone efficacy in patients with chronic kidney disease, type 2 diabetes and atherosclerotic cardiovascular disease. Eur Heart J Cardiovasc Pharmacother. 2022 Dec 15;9(1):85-93. doi: 10.1093/ehjcvp/pvac054. PMID 36251465
- [Derived] Rossing P, Burgess E, Agarwal R, Anker SD, Filippatos G, Pitt B, Ruilope LM, Gillard P, MacIsaac RJ, Wainstein J, Joseph A, Brinker M, Roessig L, Scott C, Bakris GL; FIDELIO-DKD Investigators. Finerenone in Patients With Chronic Kidney Disease and Type 2 Diabetes According to Baseline HbA1c and Insulin Use: An Analysis From the FIDELIO-DKD Study. Diabetes Care. 2022 Apr 1;45(4):888-897. doi: 10.2337/dc21-1944. PMID 35061867
- [Derived] Rossing P, Filippatos G, Agarwal R, Anker SD, Pitt B, Ruilope LM, Chan JCN, Kooy A, McCafferty K, Schernthaner G, Wanner C, Joseph A, Scheerer MF, Scott C, Bakris GL; FIDELIO-DKD Investigators. Finerenone in Predominantly Advanced CKD and Type 2 Diabetes With or Without Sodium-Glucose Cotransporter-2 Inhibitor Therapy. Kidney Int Rep. 2021 Oct 14;7(1):36-45. doi: 10.1016/j.ekir.2021.10.008. eCollection 2022 Jan. PMID 35005312
- [Derived] Agarwal R, Anker SD, Filippatos G, Pitt B, Rossing P, Ruilope LM, Boletis J, Toto R, Umpierrez GE, Wanner C, Wada T, Scott C, Joseph A, Ogbaa I, Roberts L, Scheerer MF, Bakris GL. Effects of canagliflozin versus finerenone on cardiorenal outcomes: exploratory post hoc analyses from FIDELIO-DKD compared to reported CREDENCE results. Nephrol Dial Transplant. 2022 Jun 23;37(7):1261-1269. doi: 10.1093/ndt/gfab336. PMID 34850173
- [Derived] Filippatos G, Bakris GL, Pitt B, Agarwal R, Rossing P, Ruilope LM, Butler J, Lam CSP, Kolkhof P, Roberts L, Tasto C, Joseph A, Anker SD; FIDELIO-DKD Investigators. Finerenone Reduces New-Onset Atrial Fibrillation in Patients With Chronic Kidney Disease and Type 2 Diabetes. J Am Coll Cardiol. 2021 Jul 13;78(2):142-152. doi: 10.1016/j.jacc.2021.04.079. Epub 2021 May 17. PMID 34015478
- [Derived] Erraez S, Lopez-Mesa M, Gomez-Fernandez P. Mineralcorticoid receptor blockers in chronic kidney disease. Nefrologia (Engl Ed). 2021 May-Jun;41(3):258-275. doi: 10.1016/j.nefro.2020.10.001. Epub 2020 Dec 24. English, Spanish. PMID 33358451
- [Derived] Agarwal R, Anker SD, Bakris G, Filippatos G, Pitt B, Rossing P, Ruilope L, Gebel M, Kolkhof P, Nowack C, Joseph A; FIDELIO-DKD and FIGARO-DKD Investigators. Investigating new treatment opportunities for patients with chronic kidney disease in type 2 diabetes: the role of finerenone. Nephrol Dial Transplant. 2022 May 25;37(6):1014-1023. doi: 10.1093/ndt/gfaa294. PMID 33280027
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 48 countries/regions between 17-SEP-2015 (first participant first visit) and 14-APR-2020 (last participant last visit).
Pre-assignment Details: Overall, 13911 participants were screened. Of them, 8177 participants were screening failures and 5734 participants were randomized to study treatment. 60 participants were prospectively excluded from the analyses because of Good Clinical Practice (GCP) violations, resulting in 5674 participants in the full analysis set (FAS). 16 participants did not take any study drug, resulting in 5658 participants who received study treatment.
Groups:
- Finerenone: Participants received finerenone 10 mg or 20 mg once daily in addition to standard of care therapy
Period: Overall Study
Arm/Group | Finerenone | Placebo
Started (Randomized) | 2866 | 2868
Included in FAS (60 participants were prospectively excluded from the analyses because of critical GCP violations) | 2833 | 2841
Treated | 2827 | 2831
Completed (Participants (except those with critical GCP violations) were followed up regardless of having started treatment or not, and study completion is independent of administration of study treatment. A participant included in the FAS was considered as having completed the study if there was a contact with the subject after the end-of-study (EOS) notification or if the subject died.) | 2824 | 2832
Not Completed | 42 | 36
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 4 | 6
Not completed — GCP violations | 33 | 27

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): the FAS comprised all randomized participants (except those with critical GCP violations)
Groups:
- Total: Total of all reporting groups
Arm/Group | Finerenone | Placebo | Total
Number analyzed (Participants) | 2833 | 2841 | 5674
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.44 (8.94) | 65.67 (9.16) | 65.56 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 880 | 811 | 1691
  Male | 1953 | 2030 | 3983
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 447 | 431 | 878
  Not Hispanic or Latino | 2376 | 2397 | 4773
  Unknown or Not Reported | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 78 | 76 | 154
  Asian | 717 | 723 | 1440
  Native Hawaiian or Other Pacific Islander | 11 | 7 | 18
  Black or African American | 140 | 124 | 264
  White | 1777 | 1815 | 3592
  More than one race | 101 | 86 | 187
  Unknown or Not Reported | 9 | 10 | 19
Urinary albumin-to-creatinine ratio (UACR) [Median (Inter-Quartile Range); unit: milligram/gram (mg/g)] — Population: Participants in FAS with evaluable data
  milligram/gram (mg/g)
    number analyzed (Participants) | 2831 | 2840 | 5671
    (all) | 832.72 [441.00 to 1628.14] | 867.01 [453.11 to 1644.58] | 851.87 [446.24 to 1634.22]
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Population: Participants in FAS with evaluable data
  mL/min/1.73m^2
    number analyzed (Participants) | 2832 | 2840 | 5672
    (all) | 44.36 (12.54) | 44.32 (12.57) | 44.34 (12.56)

OUTCOME MEASURES:

1. Primary Outcome: The First Occurrence of the Composite Endpoint of Onset of Kidney Failure, a Sustained Decrease of eGFR ≥40% From Baseline Over at Least 4 Weeks, or Renal Death
Description: Count of participants and time from randomization to the first occurrence of the primary renal composite outcome, onset of kidney failure, a sustained decrease of eGFR ≥40% from baseline over at least 4 weeks, or renal death were evaluated. Number of participants with the outcome event is reported as descriptive result and hazard ratio is reported as statistical analysis.
Time Frame: From randomization up until the first occurrence of the primary renal composite endpoint, or censoring at the end of the study, with an average follow-up time of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 2833 | 2841
Participants | 504 | 600
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority; p = 0.0014, Log Rank — P-value from stratified log-rank test. Significance was considered to be achieved if p-value ≤ 0.03282695; Stratified log rank test; Hazard Ratio (HR) = 0.825, 95% CI 2-sided [0.732 to 0.928] — A stratified Cox proportional hazards regression model was used to provide a point estimate of the hazard ratio and a corresponding two-sided 95% confidence interval

2. Secondary Outcome: The First Occurrence of the Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke, or Hospitalization for Heart Failure
Description: Count of participants and time from randomization to the first occurrence of the key secondary cardiovascular (CV) composite outcome, CV death, non-fatal myocardial infarction (MI), non-fatal stroke, or hospitalization for heart failure were evaluated. Number of participants with the outcome event is reported as descriptive result and hazard ratio is reported as statistical analysis.
Time Frame: From randomization up until the first occurrence of the key secondary CV composite endpoint, or censoring at the end of the study, with an average of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 2833 | 2841
Participants | 367 | 420
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority; p = 0.0339, Log Rank — P-value from stratified log-rank test. Significance was considered to be achieved if p-value ≤ 0.04967388; Stratified log rank test; Hazard Ratio (HR) = 0.860, 95% CI 2-sided [0.747 to 0.989] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: All-cause Mortality
Description: Count of participants and time from randomization until death due to any cause were evaluated. Number of participants with outcome death is reported as descriptive result and hazard ratio is reported as statistical analysis. Number of participants with outcome death reported here includes deaths occurred after randomization until the end of the study visit. Deaths after end of study visit are not included in this table.
Time Frame: From randomization up until death due to any cause, or censoring at the end of the study visit, with an average of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 2833 | 2841
Participants | 219 | 244
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — If treatment effect on both primary and key secondary endpoint is significant, other secondary efficacy endpoints (i.e. all-cause mortality, all-cause hospitalization, change in UACR from baseline to Month 4, and secondary renal composite endpoint) will be tested hierarchically, starting with all-cause mortality. If treatment effect on all-cause mortality was not significant, all other endpoints would be tested in an exploratory manner; p = 0.2348, Log Rank — P-value from stratified log-rank test. Significance was considered to be achieved if p-value ≤ 0.04967388; Stratified log rank test; Hazard Ratio (HR) = 0.895, 95% CI 2-sided [0.746 to 1.075] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: All-cause Hospitalization
Description: Count of participants and time from randomization to the first occurrence of a hospitalization event were evaluated. Number of participants with the event is reported as descriptive result and hazard ratio is reported as statistical analysis.
Time Frame: From randomization up until the first occurrence of the hospitalization due to any cause, or censoring at the end of study, with an average of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 2833 | 2841
Participants | 1263 | 1321
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1623, Log Rank — P-value from stratified log-rank test; Stratified log rank test; Hazard Ratio (HR) = 0.946, 95% CI 2-sided [0.876 to 1.022] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Urinary Albumin-to-creatinine Ratio (UACR) From Baseline to Month 4
Description: First morning void urine samples were collected to evaluate the urinary albumin-to-creatinine ratio (UACR). Month 4 was the visit closest to day 120 within a time window of 120 ± 30 days after randomization. If no measurements were available in this time window, the participant was excluded from this analysis. Ratio of UACR at Month 4 to UACR at baseline is reported as the change.
Time Frame: From baseline up until Month 4
Population: Subjects in full analysis set with measurements available within the time window of Month 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 2711 | 2705
Ratio | 0.655 [0.637 to 0.673] | 0.952 [0.927 to 0.979]
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANCOVA — P-value from F-test of equal means between the treatment groups; Ratio of least squares means = 0.688, 95% CI 2-sided [0.662 to 0.715]

6. Secondary Outcome: The First Occurrence of the Composite Endpoint of Onset of Kidney Failure, a Sustained Decrease in eGFR of ≥57% From Baseline Over at Least 4 Weeks, or Renal Death
Description: Count of participants and time from randomization to the first occurrence of the secondary renal composite outcome, onset of kidney failure, a sustained decrease in eGFR of ≥57% from baseline over at least 4 weeks, or renal death were evaluated. Number of participants with the outcome event is reported as descriptive result and hazard ratio is reported as statistical analysis.
Time Frame: From randomization up until the first occurrence of the composite primary endpoint, or censoring at the end of the study, with an average of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 2833 | 2841
Participants | 252 | 326
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0012, Log Rank — P-value from stratified log-rank test; Stratified log rank test; Hazard Ratio (HR) = 0.763, 95% CI 2-sided [0.648 to 0.900] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: After the first dose of study drug up to 3 days after any temporary or permanent interruption of study drug, with an average treatment duration of 27 months
Description: Adverse events are reported for the safety analysis set (SAF) that comprised all randomized subjects who took at least 1 dose of study drug. Adverse event reporting for the all-cause mortality considers all deaths in full analysis set (FAS, comprised all randomized participants except those with critical GCP violations) that occurred at any time during the study after randomization, including deaths after end of study visit (with an average study duration of 32 months).
Arm/Group | Finerenone | Placebo
All-Cause Mortality (participants affected / at risk) | 222/2833 | 250/2841
Serious Adverse Events (participants affected / at risk) | 902/2827 | 971/2831
Other Adverse Events (participants affected / at risk) | 1602/2827 | 1584/2831
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (N=2827) | Placebo (N=2831)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 19 (21)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (6) | 6 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (6)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 5 (5)
Aortic valve disease mixed (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 10 (10)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 8 (8)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 8 (8) | 5 (5)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 4 (4)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 2 (3)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Bifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Ischaemic mitral regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Factor VIII deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Truncus arteriosus persistent (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Goitre (Endocrine disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 2 (2)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 19 (22) | 12 (15)
Cataract diabetic (Eye disorders) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 1 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 3 (4) | 7 (8)
Ectropion (Eye disorders) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 6 (10) | 1 (1)
Lens dislocation (Eye disorders) | 1 (2) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1)
Optic disc haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 2 (2)
Retinal artery occlusion (Eye disorders) | 0 (0) | 2 (2)
Retinal detachment (Eye disorders) | 4 (7) | 2 (3)
Retinal haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 2 (2) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 6 (8) | 7 (9)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 2 (2)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 1 (1)
Tractional retinal detachment (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (5)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 6 (6)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (3) | 3 (3)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (16) | 7 (9)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Intestinal angina (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 7 (8) | 8 (8)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (6) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 5 (5) | 7 (7)
Chilaiditi's syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (3)
Chest pain (General disorders) | 13 (15) | 18 (20)
Death (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 2 (2) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 2 (2)
Generalised oedema (General disorders) | 1 (1) | 3 (3)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 4 (4) | 1 (1)
Oedema peripheral (General disorders) | 8 (10) | 7 (7)
Pyrexia (General disorders) | 4 (5) | 2 (2)
Soft tissue inflammation (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Hernia pain (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Oedema due to renal disease (General disorders) | 0 (0) | 2 (5)
Inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Device intolerance (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 4 (4)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 9 (10)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 12 (14) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 5 (5)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 3 (3)
Appendicitis perforated (Infections and infestations) | 2 (2) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 9 (9) | 13 (15)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 26 (30) | 22 (23)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 5 (5)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 3 (3)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 11 (11) | 14 (16)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 5 (5) | 5 (5)
Gastroenteritis (Infections and infestations) | 9 (9) | 13 (13)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Infected skin ulcer (Infections and infestations) | 4 (6) | 3 (3)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 7 (8) | 3 (3)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 2 (2) | 5 (5)
Localised infection (Infections and infestations) | 7 (7) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 2 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 14 (14) | 12 (12)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 70 (75) | 103 (115)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis (Infections and infestations) | 7 (7) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 5 (5) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 15 (15) | 17 (18)
Septic shock (Infections and infestations) | 3 (3) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Splenic abscess (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 21 (22) | 23 (30)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (4) | 3 (3)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 5 (5) | 7 (9)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelocystitis (Infections and infestations) | 2 (3) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (2)
Peritonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 1 (1)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 5 (5) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 3 (3) | 0 (0)
Peritoneal tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 3 (4)
Diabetic foot infection (Infections and infestations) | 4 (4) | 5 (5)
Abdominal abscess (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Borrelia infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 3 (4)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Nephritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bullous erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 (7) | 3 (4)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 9 (9)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 7 (8)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cardiac contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Biopsy kidney (Investigations) | 2 (2) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 4 (4)
Blood glucose increased (Investigations) | 2 (2) | 2 (2)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Colonoscopy (Investigations) | 2 (2) | 2 (2)
Endoscopy small intestine (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 5 (5) | 4 (4)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 3 (3)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Cardiac pacemaker evaluation (Investigations) | 1 (1) | 0 (0)
Computerised tomogram abdomen (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Light chain analysis increased (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Arteriogram (Investigations) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Cardiovascular examination (Investigations) | 0 (0) | 1 (1)
Peripheral arteriogram (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 10 (12) | 16 (18)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 12 (13) | 19 (21)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Fluid overload (Metabolism and nutrition disorders) | 7 (9) | 7 (8)
Fluid retention (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 7 (8)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (20) | 23 (26)
Hyperkalaemia (Metabolism and nutrition disorders) | 42 (45) | 12 (14)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 21 (23) | 31 (33)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (12) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 14 (16) | 22 (28)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 12 (15) | 14 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (11) | 8 (8)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (16)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 5 (5)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (3)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 4 (4)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 5 (7)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiomyofibroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alcohol induced persisting dementia (Nervous system disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Brown-Sequard syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 4 (4) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve palsies multiple (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 6 (7) | 3 (4)
Dizziness (Nervous system disorders) | 6 (6) | 10 (10)
Drop attacks (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2)
Facial paralysis (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Hemiparesis (Nervous system disorders) | 0 (0) | 3 (3)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 4 (4) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 4 (4) | 2 (2)
Radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 4 (4) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 2 (3)
Syncope (Nervous system disorders) | 12 (12) | 22 (22)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 2 (2)
Neurodegenerative disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuroglycopenia (Nervous system disorders) | 1 (2) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral vasoconstriction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral microangiopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dementia with Lewy bodies (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Secondary cerebellar degeneration (Nervous system disorders) | 0 (0) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral vascular occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hemianaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Angiopathic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (2) | 3 (4)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis ulcerative (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Glomerular vascular disorder (Renal and urinary disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 3 (3) | 4 (5)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 6 (8) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 2 (3)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 3 (3) | 9 (9)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (2) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 7 (7) | 7 (7)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (7) | 3 (3)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder cyst (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 18 (23) | 16 (19)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 8 (8) | 8 (10)
Chronic kidney disease (Renal and urinary disorders) | 12 (12) | 22 (26)
Urethral stenosis (Renal and urinary disorders) | 2 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 56 (63) | 51 (55)
Bladder outlet obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Perinephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 5 (5) | 4 (4)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 3 (3)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 10 (10)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 15 (18)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 (21) | 12 (13)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (7)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (7)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 9 (10) | 16 (19)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 13 (16) | 18 (22)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 3 (3) | 3 (3)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 3 (3)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot amputation (Surgical and medical procedures) | 1 (1) | 3 (3)
Haemodialysis (Surgical and medical procedures) | 1 (1) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 3 (4) | 6 (6)
Hysterectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 (0) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 4 (5) | 6 (7)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Metatarsal excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Myomectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Physiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pterygium operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Rhinoplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 2 (2) | 0 (0)
Tenotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 4 (5) | 4 (4)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 2 (2)
Uterine prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 1 (1) | 4 (6)
Lymphadenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Radical prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Diabetes mellitus management (Surgical and medical procedures) | 3 (3) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Continuous positive airway pressure (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephroureterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreaticosplenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Maxillofacial operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Corneal transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Bladder neck operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Urethral dilation procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Dialysis device insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 1 (1)
Foot operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Colon operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Eye operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Hydrocele operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intestinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Nail operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Wound treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 4 (5) | 12 (14)
Aneurysm repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Bowel preparation (Surgical and medical procedures) | 1 (1) | 0 (0)
Retinopexy (Surgical and medical procedures) | 0 (0) | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Internal fixation of spine (Surgical and medical procedures) | 1 (1) | 0 (0)
Bile duct stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric banding reversal (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapeutic nerve ablation (Surgical and medical procedures) | 1 (2) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Metabolic surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (4)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 2 (2) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 15 (16) | 23 (26)
Hypertensive crisis (Vascular disorders) | 4 (4) | 7 (7)
Hypotension (Vascular disorders) | 7 (7) | 5 (5)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 2 (3)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 2 (2)
Thromboangiitis obliterans (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 2 (3) | 4 (5)
Hypertensive urgency (Vascular disorders) | 4 (4) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 6 (6)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (N=2827) | Placebo (N=2831)
Anaemia (Blood and lymphatic system disorders) | 201 (218) | 177 (196)
Constipation (Gastrointestinal disorders) | 128 (146) | 162 (179)
Diarrhoea (Gastrointestinal disorders) | 183 (216) | 188 (224)
Oedema peripheral (General disorders) | 183 (216) | 303 (359)
Bronchitis (Infections and infestations) | 127 (140) | 142 (188)
Nasopharyngitis (Infections and infestations) | 241 (368) | 250 (391)
Upper respiratory tract infection (Infections and infestations) | 181 (274) | 185 (262)
Urinary tract infection (Infections and infestations) | 168 (215) | 185 (259)
Glomerular filtration rate decreased (Investigations) | 177 (225) | 130 (146)
Hyperkalaemia (Metabolism and nutrition disorders) | 422 (634) | 212 (281)
Hypoglycaemia (Metabolism and nutrition disorders) | 137 (212) | 173 (299)
Arthralgia (Musculoskeletal and connective tissue disorders) | 142 (163) | 145 (157)
Back pain (Musculoskeletal and connective tissue disorders) | 175 (187) | 170 (182)
Dizziness (Nervous system disorders) | 143 (165) | 147 (162)
Hypertension (Vascular disorders) | 200 (229) | 262 (323)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT02540993/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT02540993/SAP_001.pdf